CLINICAL TRIAL: NCT03661242
Title: Integration of Exercise Into Cancer Care: A Shared Care Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Landspitali University Hospital (Other)
Collaborators: Gundersen Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: LSH-18-001
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2018-08

CONDITIONS: Cancer
Keywords: Physical activity; Exercise; Adjuvant chemotherapy
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The design is a quasi-experimental prospective double- cohort study in which a lead-in group will be enrolled and receive standard of care and an intervention group will be enrolled one year after the last lead-in patient is accrued. The intervention group will receive shared care with an oncologist and an exercise physiologist trained in providing activity and exercise guidelines to the cancer patient population.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): No intervention
- Shared care (Active Comparator): Clinic visit with Clincal Exercise Physiologist or physical therapist who does assessment and prescripes individulized physical activity plan
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — Patients in shared care arm has regular combined visits with Oncologist and Clincal Exercise Physiologist (CEP). Individual physical activity plan developed by CEP for patients in shared care arm.
  Arms: Shared care

SUMMARY:
Multiple organizations endorse physical activity for cancer patients; however the structure for oncologist prescribed exercise has not been clearly established. A focus group study previously conducted at Gundersen Health System identified a patient preference for integrated care surrounding physical activity. Thus, the focus of this study will be to investigate the effects of a shared care model on the physical activity levels of cancer patients. The shared care model will consist of regularly scheduled visits with the patient's oncologist in combination with a clinical exercise physiologist. The clinical exercise physiologist (CEP) will assist in developing an individual activity plan with the patient. The Investigators predict the shared care model patients will have a higher level of activity, functional capacity and quality of life.

DETAILED DESCRIPTION:
Numerous organizations, including the American Cancer Society, American College of Sports Medicine, National Comprehensive Cancer Network, U.S. Department of Health and Human Resources and Oncology Nursing Society have endorsed physical activity for cancer patients both when undergoing treatment and during the survivorship phase of care. Previous studies have consistently found physical activity to be associated with improved quality of life. However, current guidelines for oncologist prescribed exercise are vague and not supported with adequate training and/or education.

A focus group study previously conducted at Gundersen Health System found that oncologists' reluctance to discuss physical activity with patients is rooted in their own ability to safely guide patients through an exercise program. Cancer patients have also reported uncertainty about what types, frequency and intensity of physical activity in which to engage and it has been suggested that a referral process is critical to inclusion of exercise prescription into cancer care. Investigator´s previous study, along with others, have found that patients want advice and support about exercise while enduring the physiological and psychological side effects of treatment, yet do not want to be referred elsewhere. Thus, it seems there is a dilemma of translating safe and sustainable physical activity into standard cancer care.

A potential solution to this perceived shortcoming is a shared care model of cancer care delivery, wherein an oncologist is partnered with a certified exercise physiologist or physical therapist to develop an individualized, holistic care plan for each patient. In addition to providing the patient with standard of care cancer therapy as prescribed by the oncologist, the shared care model will also provide the patient with a customized physical activity plan developed by the exercise physiologist in consultation with the oncology staff and after meeting with the patient during a regularly scheduled oncology office visit. In this study the Investigators propose to investigate the impact of shared care visits with an oncologist and exercise physiologist on quality of life and functional capacity during cancer treatment. This model provides patients with easy access to the advice and support they desire without the need for additional referrals and travel, while ensuring a comprehensive assessment of risks and the development of safe progression of activities. Plan is to recruit total of 120 patients.

Statistical analysis will utilized a mix of descriptive and comparative statistics. Descriptive metrics will include means and associated 95% confidence intervals, medians and frequency counts. Comparison of demographic and clinical factors between study groups will utilize the Chi-square test for categorical data, the Wilcoxon rank sum test or Kruskal-Wallis test for ordinal discrete or non-normally distributed continuous data and Student's t-test or ANOVA for normally distributed continuous data. Evaluation of the primary outcome will utilize repeated measures ANOVA to compare the change overall quality of life over the study period, assessed via the FACT-G instrument, between the study groups. A p-value < 0.05 will be used as the threshold for statistical significance for all tests.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Pathologic confirmed cancer diagnosis
* Patients receiving adjuvant treatment (chemotherapy and/or radiation) with curative intent
* ECOG performance status 0-2

Exclusion Criteria:

* Unable to ambulate
* Comorbidity contraindicated PA as per treating physician
* Non-English speaker
* Receiving maintenance chemotherapy
* Breast cancer diagnosis
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy - General (FACT-G QOL) measurement. | Month 0 (first visit), month 1, month 3, month 6, month 9, month 12
  Change in score of FACT-G QOL measurement.

SECONDARY OUTCOMES:
6-minute walk test | Month 0 (first visit), month 1, month 3, month 6, month 9, month 12
  Change in 6-minute walk test
International Physical Activity Questionnaire (IPAQ) score | Month 0 (first visit), month 1, month 3, month 6, month 9, month 12
  Change in International Physical Activity Questionnaire (IPAQ) score
Patient Health Questionnaire 9 (PHQ-9) score | Month 0 (first visit), month 1, month 3, month 6, month 9, month 12
  Change in Patient Health Questionnaire (PHQ) score

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Smaradottir, MD, Principal Investigator — Landspitali University Hospital
Locations (2):
- Gundersen Health System, La Crosse, Wisconsin, United States
- Landspitali - The National University Hospital of Iceland, Reykjavik, Iceland